CLINICAL TRIAL: NCT00792948
Title: Phase II Study of Combination of Hyper-CVAD and Dasatinib (NSC-732517) With or Without Allogeneic Stem Cell Transplant in Patients With Philadelphia (Ph) Chromosome Positive and/or BCR-ABL Positive Acute Lymphoblastic Leukemia (ALL) (A BMT Study)
Brief Title: Combination Chemotherapy With or Without Donor Stem Cell Transplant in Treating Patients With Acute Lymphoblastic Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00800; NCI-2009-00800 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S0805; CDR0000624250; S0805 (Other: SWOG); S0805 (Other: CTEP); U10CA180888 (NIH); U10CA032102 (NIH)
Record Dates: First submitted 2008-11-16; First posted 2008-11-18 (Estimated); Results first posted 2017-04-26 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-08

CONDITIONS: Acute Lymphoblastic Leukemia; Adult B Acute Lymphoblastic Leukemia; Adult B Acute Lymphoblastic Leukemia With t(9;22)(q34.1;q11.2); BCR-ABL1; Adult L1 Acute Lymphoblastic Leukemia; Adult L2 Acute Lymphoblastic Leukemia; Adult T Acute Lymphoblastic Leukemia; Recurrent Adult Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Stem Cell Transplantation; Cyclophosphamide; Cytarabine; Dasatinib; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Doxorubicin; Etoposide; Filgrastim; Granulocyte Colony-Stimulating Factor; Leucovorin; Methotrexate; merphos; Methylprednisolone; exifone; Medrol Veriderm; Peripheral Blood Stem Cell Transplantation; Prednisone; deltacortene; prednylidene; Sirolimus; Tacrolimus; Whole-Body Irradiation; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (chemotherapy, transplant, maintenance) (Experimental): See Detailed Description
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dasatinib; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Biological: Filgrastim; Other: Laboratory Biomarker Analysis; Drug: Leucovorin Calcium; Drug: Methotrexate; Drug: Methylprednisolone; Procedure: Peripheral Blood Stem Cell Transplantation; Drug: Prednisone; Drug: Sirolimus; Drug: Tacrolimus; Radiation: Total-Body Irradiation; Drug: Vincristine Sulfate

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic stem cell transplant
  Other Names: Allogeneic; Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Cytarabine — Given IT
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Dasatinib — Given PO
  Other Names: BMS 354825; BMS-354825; BMS354825; Dasatinib Hydrate; Dasatinib Monohydrate; Sprycel
Drug: Dexamethasone — Given IV or PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; LenaDex; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Biological: Filgrastim — Given SC
  Other Names: Filgrastim Biosimilar Filgrastim-sndz; Filgrastim Biosimilar Tbo-filgrastim; Filgrastim XM02; Filgrastim-aafi; Filgrastim-ayow; Filgrastim-sndz; G-CSF; Granix; Neupogen; Neutroval; Nivestim; Nivestym; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; Releuko; rG-CSF; Tbo-filgrastim; Tevagrastim; XM02; Zarxio
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Drug: Methotrexate — Given IV or IT
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Jylamvo; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Methylprednisolone — Given IV
  Other Names: Adlone; Caberdelta M; DepMedalone; Depo Moderin; Depo-Nisolone; Duralone; Emmetipi; Esametone; Firmacort; Medlone 21; Medrate; Medrol; Medrol Veriderm; Medrone; Mega-Star; Meprolone; Methylprednisolonum; Metilbetasone Solubile; Metrocort; Metypresol; Metysolon; Predni-M-Tablinen; Prednilen; Radilem; Sieropresol; Solpredone; Summicort; Urbason; Veriderm Medrol; Wyacort
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo allogeneic stem cell transplant
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood; Peripheral Blood Progenitor Cell Transplantation; PERIPHERAL BLOOD STEM CELL TRANSPLANT; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Drug: Sirolimus — Given PO
  Other Names: AY 22989; AY-22989; AY22989; RAPA; Rapamune; Rapamycin; SILA 9268A; SILA-9268A; SILA9268A; WY 090217; WY-090217; WY090217
Drug: Tacrolimus — Given IV
  Other Names: FK 506; FK-506; FK506; Fujimycin; Hecoria; Prograf; Protopic; Tacforius
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: SCT_TBI; TBI; Total Body Irradiation; Whole Body; Whole Body Irradiation; Whole-Body Irradiation
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase II trial is studying the side effects of giving combination chemotherapy together with or without donor stem cell transplant and to see how well it works in treating patients with acute lymphoblastic leukemia. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells. Giving chemotherapy and total-body irradiation before a donor stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test whether the relapse-free survival after allogeneic stem cell transplantation among Philadelphia chromosome positive and/or breakpoint cluster region (BCR)/Abelson murine leukemia viral oncogene (ABL) positive acute lymphoblastic leukemia (ALL) patients given an intensive short-term chemotherapy regimen of fractionated cyclophosphamide, vincristine sulfate, doxorubicin hydrochloride, and dexamethasone (hyper-CVAD) in combination with the tyrosine kinase inhibitor dasatinib is sufficiently high to warrant further investigation.

SECONDARY OBJECTIVES:

I. To test whether the continuous complete remission rate for previously untreated Philadelphia chromosome positive and/or BCR/ABL positive acute lymphoblastic leukemia (ALL) patients given an intensive short-term chemotherapy regimen of hyper-CVAD in combination with the tyrosine kinase inhibitor dasatinib is sufficiently high to warrant phase III investigation.

II. To investigate in a preliminary manner the relative effectiveness of minimal residual disease (MRD) detection using real-time quantitative polymerase chain reaction (PCR) for BCR/ABL versus flow cytometry to predict the outcome of patients treated by the hyper-CVAD + dasatinib regimen and/or allogeneic stem cell transplant.

TERTIARY OBJECTIVES:

I. To estimate the frequency and severity of toxicities of the intensive short-term chemotherapy regimen in these patients.

II. To estimate the overall survival of all patients on this study.

OUTLINE:

INDUCTION/CONSOLIDATION THERAPY: All patients receive both of the following regimens in alternating courses:

COURSES 1, 3, 5, 7 or 3, 5, 7, 9: Patients receive cyclophosphamide intravenously (IV) over 3 hours twice daily (BID) on days 1-3; doxorubicin hydrochloride IV over 24 hours on day 4; vincristine sulfate IV over 30 minutes on days 4 and 11; dexamethasone IV or orally (PO) once daily (QD) on days 1-4 and 11-14; dasatinib PO QD on days 1-14; cytarabine intrathecally (IT) on day 7; methotrexate IT on day 2; and filgrastim (G-CSF) subcutaneously (SC) QD or BID.

COURSES 2, 4, 6, 8: Patients receive high-dose methotrexate IV over 24 hours on day 1; methylprednisolone IV over 30 minutes BID on days 1-3; dasatinib PO QD on days 1-14; high-dose cytarabine IV over 2 hours BID on days 2-3; leucovorin calcium IV on days 2 or 3; methotrexate IT on day 2; cytarabine IT on day 7; and G-CSF SC QD or BID.

Treatment repeats every 14-21 days for 8 courses in the absence of disease progression, unacceptable toxicity, or if patient achieves complete remission (CR) or complete remission with incomplete platelet recovery (CRi).

MAINTENANCE THERAPY*: Patients receive vincristine sulfate IV over 30 minutes on day 1, prednisone PO QD on days 1-5, and dasatinib PO QD on days 1-28.

Treatment repeats every month for 24 courses in the absence of disease progression or unacceptable toxicity or until the transplant is ready.

INTENSIFICATION: For courses 6 and 13, patients receive cyclophosphamide IV over 3 hours BID on days 1-3; doxorubicin hydrochloride IV over 24 hours on day 4; vincristine sulfate IV over 30 minutes on days 4 and 11; dexamethasone IV or PO QD on days 1-4 and 11-14; dasatinib PO QD on days 1-14; and G-CSF SC QD or BID.

NOTE: *Only if transplantation is not ready after induction/consolidation therapy or patients are not undergoing a transplant.

ALLOGENEIC STEM CELL TRANSPLANTATION (FOR PATIENTS ACHIEVING CR OR CRi):

CONDITIONING REGIMEN: Patients receive 1 of the following regimens:

REGIMEN A: Patients receive total-body irradiation (TBI) QD on days -7 to -4 and cyclophosphamide IV on days -3 and -2.

REGIMEN B: Patients receive TBI BID on days -6 to -4 and cyclophosphamide IV on days -3 and -2.

REGIMEN C: Patients receive cyclophosphamide IV on days -7 and -6 and TBI QD on days -4 to -1.

REGIMEN D: Patients receive cyclophosphamide IV on days -6 and -5 and TBI BID on days -3 to -1.

REGIMEN E: Patients receive TBI QD on days -7 to -4 and etoposide IV on day -3.

REGIMEN F: Patients receive TBI BID on days -6 to -4 and etoposide IV on day -3.

ALLOGENEIC STEM CALL TRANSPLANTATION: Patients undergo allogeneic stem cell transplantation on day 0.

GRAFT-VS-HOST DISEASE (GVHD) PROPHYLAXIS: Patients receive 1 of the following regimens:

REGIMEN A: Patients receive sirolimus PO and tacrolimus IV continuously (changing to PO BID) beginning on day -3 and continuing for 6 months.

REGIMEN B: Patients receive tacrolimus IV continuously (changing to PO BID) and continuing for 6 months, and methotrexate IV on days 1, 3, 6, and 11.

SINGLE-AGENT THERAPY: After completion of maintenance therapy or beginning on day 100 post-transplantation, patients receive dasatinib PO QD for up to 5 years.

After completion of study therapy, patients are followed every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* INDUCTION/CONSOLIDATION REGISTRATION:
* Patients must have a morphologic diagnosis of acute lymphoblastic leukemia (ALL), with evidence of ALL involvement in bone marrow and/or blood; patients with only extramedullary disease in the absence of bone marrow or blood involvement are not eligible; patients with M0 acute myeloid leukemia (AML) or mixed lineage leukemia are not eligible for this study; patients with L3 (Burkitts) are also not eligible

  * For ALL in marrow or peripheral blood, immunophenotyping of the blood or marrow lymphoblasts must be performed to determine lineage (B cell, T-cell, or mixed B/T cell); NOTE: appropriate marker studies including cluster of differentiation (CD)19 (B cell), CD10, CD5, and CD7 (T cell) must be performed; co-expression of myeloid antigens (CD13 and CD33) will not exclude patients; if possible, the lineage specific markers cytoplasmic CD22 or CD79a (B cells), cytoplasmic CD3 (T cells) and cytoplasmic myeloperoxidase (MPO) (myeloid cells) must be determined
* Patients may have received no more than one course of remission induction therapy for ALL; patients who have received any post-remission therapy for ALL or who have relapsed from complete remission are not eligible; (patients with previously untreated ALL can be eligible, and patients who have received one course of remission induction therapy for ALL can be eligible, regardless of their response to therapy); patients may have received no more than 14 days of tyrosine kinase inhibitor therapy prior to registration; any prior induction chemotherapy must have been completed no more than 28 days prior to registration

  * NOTE: If the patient has been initiated on the protocol defined regimen (i.e. the hyper-CVAD regimen without a tyrosine kinase inhibitor) before the Philadelphia chromosome (Ph)/BCR-ABL status was known, the patient may be registered on the protocol and start dasatinib; in this first course, dasatinib will be administered up to day 14 (i.e. if the patient is registered on day 5 and starts therapy on day 6, only 8 days of dasatinib will be administered and dasatinib will be completed on day 14)
* For patients who have received any prior therapy that was NOT remission induction therapy, one of the following must be true:

  * At least 6 weeks must have elapsed since any monoclonal antibodies were given, at least 7 days must have elapsed since any other treatment was given, and all toxicities of the remission induction therapy must have resolved to grade =< 2
  * The patient must have rapidly progressive disease (per institutional guidelines)
* For previously treated patients, the study chair must be contacted before registration, in order to determine the regimen to be given in the first course of induction/consolidation therapy, based on prior therapy
* Patients must be Philadelphia (Ph) positive and/or BCR/ABL positive as confirmed by standard cytogenetics, fluorescent in situ hybridization (FISH), and/or polymerase chain reaction (PCR) testing performed by local laboratory; NOTE: samples will be submitted centrally for verification of results
* Patients must have a bilirubin =< 3.0 x institutional upper limit of normal (IULN) within 14 days prior to registration
* Patients must have serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 3.0 x IULN and/or serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 3.0 x IULN within 14 days prior to registration; if both tests are done then both values must be =< 3.0 x IULN
* Patients must have a serum creatinine =< 3.0 x IULN within 14 days prior to registration
* Patients must not have active pericardial effusion, ascites, or pleural effusion of any grade; exception: if the effusion is suspected to be related to the leukemia, the patient may have pericardial effusion of =< grade 2 or pleural effusion =< grade 1
* Patients may not have any clinically significant cardiovascular disease including the following:

  * Myocardial infarction or ventricular tachyarrhythmia within 6 months
  * Prolonged corrected QT (QTc) >= 480 msec (Fridericia correction)
  * Ejection fraction less than institutional normal
  * Major conduction abnormality (unless a cardiac pacemaker is present)
  * Patients with any cardiopulmonary symptoms of unknown cause (e.g. shortness of breath, chest pain, etc.) should be evaluated by a baseline echocardiogram with or without stress test as needed in addition to electrocardiogram (EKG) to rule out QTc prolongation; the patient may be referred to a cardiologist at the discretion of the principal investigator; patients with underlying cardiopulmonary dysfunction should be excluded from the study
* Patients must have Zubrod performance status of 0-2
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years
* Collection and submission of pre-treatment cytogenetic specimens must be completed within 28 days prior to registration on S0805
* Collection and submission of pretreatment marrow and/or peripheral blood specimens for cellular and molecular studies, including verification of BCR/ABL status must be completed within 28 days prior to registration
* Patients must not be pregnant or nursing; women/men of reproductive potential must have agreed to use an effective contraceptive method; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* Patients must not have prior history of known type I hypersensitivity or anaphylactic reactions to doxorubicin
* Patients or their legally authorized representative must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* At the time of patient registration, the treating institution's name and identification (ID) number must be provided to the Data Operations Center in Seattle in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered into the data base
* MAINTENANCE/INTENSIFICATION:
* Patient must have achieved CR or CRi within 2 courses of Induction/Consolidation Chemotherapy; patient must remain in CR or CRi until beginning Maintenance Chemotherapy and this must be re-documented by bone marrow and peripheral blood examination within 28 days prior to registration to Step 2
* All treatment related toxicities must have resolved to =< grade 2
* Patients must not have received allogeneic stem cell transplant
* TRANSPLANT REGISTRATION:
* Patients must have an available completely matched sibling donor or a 10/10 matched non-sibling donor
* Patients must have allogeneic stem cell transplant arranged prior to registration to Step 3
* Patients must have documented CR or CRi within 14 days prior to registration to Step 3
* Patients must not be HIV + (human immunodeficiency virus); a negative HIV test must be obtained within 14 days prior to registration
* POST TRANSPLANT/POST-MAINTENANCE SINGLE-AGENT DASATINIB THERAPY:
* Patients must have reached day 100 post transplant or must have completed protocol maintenance/intensification (or must have been approved by the Study Chair after early removal from maintenance/intensification)
* Patients must be in CR or CRi based on bone marrow and peripheral blood examination within 28 days prior to registration to Step 4
* Patients must have recovered to =< grade 2 from all treatment related toxicity

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2026-01-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Ravandi-Kashani, Principal Investigator — SWOG Cancer Research Network
Locations (157):
- United States (157):
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - MacNeal Hospital and Cancer Center, Berwyn, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - DuPage Medical Group-Ogden, Naperville, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Reid Health, Richmond, Indiana
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - HaysMed, Hays, Kansas
  - Hutchinson Regional Medical Center, Hutchinson, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Hematology/Oncology Clinic PLLC, Baton Rouge, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University Health Truman Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - The Jewish Hospital, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Clinton Memorial Hospital/Foster J Boyd Regional Cancer Center, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Statler A, Othus M, Erba HP, Chauncey TR, Radich JP, Coutre S, Advani A, Nand S, Ravandi F, Mukherjee S, Sekeres MA. Comparable outcomes of patients eligible vs ineligible for SWOG leukemia studies. Blood. 2018 Jun 21;131(25):2782-2788. doi: 10.1182/blood-2018-01-826693. Epub 2018 Apr 4. PMID 29618479

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: See Detailed Description
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo allogeneic stem cell transplant
  Cyclophosphamide: Given IV
  Cytarabine: Given IT
  Dasatinib: Given PO
  Dexamethasone: Given IV or PO
  Doxorubicin Hydrochloride: Given IV
  Etoposide: Given IV
  Filgrastim: Given SC
  Laboratory Biomarker Analysis: Correlative studies
  Leucovorin Calcium: Given IV
  Methotrexate: Given IV or IT
  Methylprednisolone: Given IV
  Peripheral Blood Stem Cell Transplantation: Undergo allogeneic stem cell transplant
  Prednisone: Given PO
  Sirolimus: Given PO
  Tacrolimus: Given IV
  Total-Body Irradiation: Undergo TBI
  Vincristine Sulfate: Given IV
Period: Overall Study
Arm/Group | Treatment
Started | 97 (Patients registered to induction/consolidation step)
Completed | 69 (Patients who completed induction/consolidation step)
Not Completed | 28
Not completed — Adverse Event | 6
Not completed — Death | 4
Not completed — Withdrawal by Subject | 3
Not completed — Ineligible | 2
Not completed — Insurance denial - not treated | 1
Not completed — Physician Decision | 11
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Analysis includes eligible patients who received treatment.
Arm/Group | Treatment
Number analyzed (Participants) | 94
Age, Continuous [Median (Full Range); unit: years] | 44 [20.5 to 60.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 42

OUTCOME MEASURES:

1. Primary Outcome: Relapse-free Survival (RFS) After Allogeneic Stem Cell Transplantation
Description: Will be estimated using the method of Kaplan-Meier.
Time Frame: 12 months
Population: Patients who received allogeneic stem cell transplant
Measure: Number (95% Confidence Interval); unit: Probability of 12-month RFS
Arm/Group | Treatment
Number analyzed (Participants) | 40
Probability of 12-month RFS | 0.83 [0.67 to 0.91]

2. Secondary Outcome: Continuous Complete Remission (CCR) Rate
Description: Will be testing using an exact binomial test
Time Frame: 18 months
Population: Patients who had not received prior ALL therapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 60
percentage of participants | 57 [43 to 69]

3. Other Pre Specified Outcome: Overall Survival (OS)
Description: OS will be estimated using the method of Kaplan-Meier.
Time Frame: From the date of initial registration on the study until death from any cause, assessed up to 5 years
Population: Analysis includes eligible patients who received treatment.
Measure: Number (95% Confidence Interval); unit: Probability of surviving 12 months
Arm/Group | Treatment
Number analyzed (Participants) | 94
Probability of surviving 12 months | 0.88 [0.80 to 0.93]

4. Other Pre Specified Outcome: MRD as Assessed Using Real-time Quantitative Polymerase Chain Reaction and Flow Cytometry
Description: Correlation between the two measures of MRD measured on the same remission specimens will be examined using scatterplots and correlation analysis. The prognostic effect for relapse of each measure will be illustrated using cumulative incidence plots, and estimated using Cox regression models. This outcome will be reported as funding allows.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: Analysis includes eligible patients who were assessed for adverse events.
Groups:
- Induction/Consolidation: Patients receive up to 8 courses, alternating between hyper-CVAD plus dasatinib and high dose methotrexate and cytarabine plus dasatinib. There are nine possible induction/consolidation courses.
- Vincristine/Prednisone/Dasatinib: Patients receive vincristine IV on day 1, prednisone PO on days 1 to 5, and dasatinib PO on days 1 to 28 for up to 24 courses or until transplant is available.
- Allogeneic Stem Cell Transplant: Patients who have an available sibling donor or a 10/10 matched unrelated donor will be removed from therapy and proceed directly to allogeneic stem cell transplant after achieving CR or CRi.
- Dasatinib: Patients receive Single-Agent Dasatinib therapy PO every day for up to five years from original registration.
Arm/Group | Induction/Consolidation | Vincristine/Prednisone/Dasatinib | Allogeneic Stem Cell Transplant | Dasatinib
Serious Adverse Events (participants affected / at risk) | 43/93 | 5/22 | 2/4 | 10/39
Other Adverse Events (participants affected / at risk) | 89/93 | 22/22 | 0/4 | 36/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction/Consolidation (N=93) | Vincristine/Prednisone/Dasatinib (N=22) | Allogeneic Stem Cell Transplant (N=4) | Dasatinib (N=39)
Febrile neutropenia (Blood and lymphatic system disorders) | 26 | 1 | 0 | 0
Hemoglobin (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1
SVT and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
SVT and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Enteritis (inflammation of the small bowel) (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal-Other (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Pain - Abdomen NOS (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Perforation, GI - Stomach (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Edema: limb (General disorders) | 0 | 1 | 0 | 0
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 | 1 | 0 | 0
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 1 | 0 | 0 | 1
Pain - Chest/thorax NOS (General disorders) | 0 | 1 | 0 | 0
Sudden death (General disorders) | 1 | 0 | 0 | 0
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 | 1 | 0 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Blood (Infections and infestations) | 5 | 0 | 0 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Catheter-rel (Infections and infestations) | 1 | 0 | 0 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Lung (Infections and infestations) | 1 | 0 | 0 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Skin (Infections and infestations) | 2 | 0 | 0 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Upper airway (Infections and infestations) | 1 | 1 | 0 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Catheter (Infections and infestations) | 1 | 0 | 0 | 0
Infection with unknown ANC - Blood (Infections and infestations) | 8 | 1 | 0 | 0
Infection with unknown ANC - Bronchus (Infections and infestations) | 1 | 0 | 0 | 0
Infection with unknown ANC - Catheter-related (Infections and infestations) | 3 | 0 | 0 | 0
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 5 | 1 | 0 | 0
Infection with unknown ANC - Meninges (meningitis) (Infections and infestations) | 0 | 0 | 0 | 1
Infection with unknown ANC - Scrotum (Infections and infestations) | 0 | 1 | 0 | 0
Infection with unknown ANC - Sinus (Infections and infestations) | 1 | 0 | 0 | 0
Infection with unknown ANC - Skin (cellulitis) (Infections and infestations) | 2 | 0 | 0 | 0
Infection with unknown ANC - Soft tissue NOS (Infections and infestations) | 1 | 0 | 0 | 0
Infection-Other (Infections and infestations) | 5 | 1 | 1 | 3
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 5 | 0 | 0 | 0
AST, SGOT (Investigations) | 2 | 1 | 0 | 0
Alkaline phosphatase (Investigations) | 0 | 1 | 0 | 0
Bilirubin (hyperbilirubinemia) (Investigations) | 1 | 0 | 0 | 0
Carbon monoxide diffusion capacity (DL(co)) (Investigations) | 1 | 0 | 1 | 1
Creatinine (Investigations) | 2 | 0 | 0 | 0
GGT (gamma-glutamyl transpeptidase) (Investigations) | 1 | 0 | 0 | 0
Leukocytes (total WBC) (Investigations) | 2 | 0 | 0 | 0
Lymphopenia (Investigations) | 2 | 0 | 0 | 0
Metabolic/Laboratory-Other (Investigations) | 1 | 0 | 0 | 0
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 7 | 0 | 0 | 0
Platelets (Investigations) | 5 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0
Muscle weakness, not d/t neuropathy - Extrem-lower (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain - Back (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain - Joint (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Soft tissue necrosis - Extremity-lower (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Secondary Malignancy-poss rel to cancer Tx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Muscle weakness, not d/t neuropathy - Facial (Nervous system disorders) | 0 | 0 | 0 | 1
Neurology-Other (Nervous system disorders) | 1 | 0 | 0 | 0
Neuropathy: motor (Nervous system disorders) | 1 | 0 | 0 | 0
Pain - Head/headache (Nervous system disorders) | 2 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1
Confusion (Psychiatric disorders) | 1 | 0 | 0 | 0
Mood alteration - anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 0 | 1 | 0 | 0
Hemorrhage, GU - Urinary NOS (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 2 | 0 | 0 | 1
Adult respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Carbon monoxide diffusion capacity (DL(co)) (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary/Upper Respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Petechiae/purpura (hemorrhage into skin or mucosa) (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hematoma (Vascular disorders) | 1 | 0 | 0 | 1
Hemorrhage/Bleeding-Other (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Induction/Consolidation (N=93) | Vincristine/Prednisone/Dasatinib (N=22) | Allogeneic Stem Cell Transplant (N=4) | Dasatinib (N=39)
Blood/Bone Marrow-Other (Blood and lymphatic system disorders) | 5 | 1 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 28 | 1 | 0 | 1
Hemoglobin (Blood and lymphatic system disorders) | 69 | 14 | 0 | 29
Lymphatics-Other (Blood and lymphatic system disorders) | 5 | 0 | 0 | 3
Cardiac General-Other (Cardiac disorders) | 3 | 0 | 0 | 2
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 | 0 | 0 | 5
SVT and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 11 | 0 | 0 | 2
Cushingoid appearance (Endocrine disorders) | 0 | 0 | 0 | 2
Cataract (Eye disorders) | 0 | 0 | 0 | 3
Dry eye syndrome (Eye disorders) | 2 | 0 | 0 | 12
Ocular/Visual-Other (Eye disorders) | 6 | 4 | 0 | 4
Pain - Eye (Eye disorders) | 7 | 0 | 0 | 1
Vision-blurred vision (Eye disorders) | 5 | 6 | 0 | 5
Colitis (Gastrointestinal disorders) | 1 | 1 | 0 | 3
Constipation (Gastrointestinal disorders) | 41 | 10 | 0 | 10
Diarrhea (Gastrointestinal disorders) | 39 | 6 | 0 | 22
Distention/bloating, abdominal (Gastrointestinal disorders) | 9 | 1 | 0 | 2
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 | 0 | 0 | 7
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Gastrointestinal-Other (Gastrointestinal disorders) | 4 | 2 | 0 | 5
Heartburn/dyspepsia (Gastrointestinal disorders) | 22 | 3 | 0 | 7
Hemorrhoids (Gastrointestinal disorders) | 12 | 1 | 0 | 1
Malabsorption (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 15 | 1 | 0 | 3
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 17 | 1 | 0 | 2
Nausea (Gastrointestinal disorders) | 78 | 11 | 0 | 28
Pain - Abdomen NOS (Gastrointestinal disorders) | 33 | 6 | 0 | 10
Pain - Oral cavity (Gastrointestinal disorders) | 7 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 51 | 5 | 0 | 23
Edema: head and neck (General disorders) | 10 | 2 | 0 | 5
Edema: limb (General disorders) | 31 | 7 | 0 | 21
Edema: trunk/genital (General disorders) | 1 | 0 | 0 | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 59 | 11 | 0 | 27
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 30 | 7 | 0 | 11
Flu-like syndrome (General disorders) | 0 | 0 | 0 | 5
Injection site reaction/extravasation changes (General disorders) | 4 | 0 | 0 | 2
Pain - Chest/thorax NOS (General disorders) | 5 | 3 | 0 | 4
Pain - Pain NOS (General disorders) | 1 | 0 | 0 | 4
Pain-Other (General disorders) | 10 | 3 | 0 | 9
Rigors/chills (General disorders) | 9 | 3 | 0 | 7
Syndromes-Other (General disorders) | 1 | 0 | 0 | 3
Allergic reaction/hypersensitivity (Immune system disorders) | 9 | 2 | 0 | 5
Allergy/Immunology-Other (Immune system disorders) | 3 | 0 | 0 | 3
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 5 | 3 | 0 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Blood (Infections and infestations) | 12 | 0 | 0 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Lung (Infections and infestations) | 7 | 0 | 0 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Oral cav-gums (Infections and infestations) | 5 | 0 | 0 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Blood (Infections and infestations) | 1 | 1 | 0 | 2
Inf w/normal ANC or Gr 1-2 neutrophils - Bronchus (Infections and infestations) | 1 | 1 | 0 | 2
Inf w/normal ANC or Gr 1-2 neutrophils - Eye NOS (Infections and infestations) | 0 | 0 | 0 | 2
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 7 | 2 | 0 | 4
Inf w/normal ANC or Gr 1-2 neutrophils - Sinus (Infections and infestations) | 1 | 1 | 0 | 6
Inf w/normal ANC or Gr 1-2 neutrophils - Skin (Infections and infestations) | 4 | 0 | 0 | 4
Inf w/normal ANC or Gr 1-2 neutrophils - UTI (Infections and infestations) | 2 | 1 | 0 | 4
Inf w/normal ANC or Gr 1-2 neutrophils - Up airway (Infections and infestations) | 6 | 1 | 0 | 9
Inf w/unknown ANC - Middle ear (otitis media) (Infections and infestations) | 0 | 0 | 0 | 2
Infection with unknown ANC - Upper airway NOS (Infections and infestations) | 0 | 1 | 0 | 3
Infection with unknown ANC - Urinary tract NOS (Infections and infestations) | 1 | 0 | 0 | 2
Infection-Other (Infections and infestations) | 10 | 6 | 0 | 7
Bruising (in absence of Gr 3-4 thrombocytopenia) (Injury, poisoning and procedural complications) | 8 | 3 | 0 | 7
Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 44 | 12 | 0 | 21
AST, SGOT (Investigations) | 46 | 12 | 0 | 18
Alkaline phosphatase (Investigations) | 27 | 4 | 0 | 12
Bilirubin (hyperbilirubinemia) (Investigations) | 27 | 0 | 0 | 5
Cholesterol, serum-high (hypercholesterolemia) (Investigations) | 0 | 3 | 0 | 5
Creatinine (Investigations) | 19 | 4 | 0 | 18
Fibrinogen (Investigations) | 8 | 0 | 0 | 0
INR (of prothrombin time) (Investigations) | 8 | 1 | 0 | 2
Leukocytes (total WBC) (Investigations) | 60 | 15 | 0 | 19
Lymphopenia (Investigations) | 40 | 5 | 0 | 17
Metabolic/Laboratory-Other (Investigations) | 12 | 2 | 0 | 5
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 56 | 9 | 0 | 20
PTT (Partial thromboplastin time) (Investigations) | 6 | 1 | 0 | 0
Platelets (Investigations) | 66 | 11 | 0 | 19
Weight gain (Investigations) | 9 | 2 | 0 | 6
Weight loss (Investigations) | 13 | 0 | 0 | 9
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 40 | 5 | 0 | 12
Anorexia (Metabolism and nutrition disorders) | 34 | 3 | 0 | 14
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 6 | 0 | 0 | 2
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 49 | 8 | 0 | 16
Dehydration (Metabolism and nutrition disorders) | 7 | 1 | 0 | 5
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 54 | 8 | 0 | 14
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 9 | 2 | 0 | 5
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 13 | 1 | 0 | 1
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 23 | 3 | 0 | 11
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 17 | 1 | 0 | 8
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 8 | 1 | 0 | 6
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 58 | 8 | 0 | 12
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 9 | 3 | 0 | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 27 | 5 | 0 | 9
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 3 | 2 | 0 | 4
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 6 | 0 | 0 | 5
Joint-function (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Muscle weakness, not d/t neuropathy - Extrem-lower (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0 | 4
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 10 | 4 | 0 | 3
Musculoskeletal/Soft Tissue-Other (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0 | 6
Pain - Back (Musculoskeletal and connective tissue disorders) | 26 | 6 | 0 | 8
Pain - Bone (Musculoskeletal and connective tissue disorders) | 17 | 1 | 0 | 5
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 5 | 0 | 0 | 4
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 10 | 2 | 0 | 12
Pain - Joint (Musculoskeletal and connective tissue disorders) | 7 | 2 | 0 | 13
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 16 | 3 | 0 | 13
Pain - Neck (Musculoskeletal and connective tissue disorders) | 7 | 3 | 0 | 4
Dizziness (Nervous system disorders) | 22 | 4 | 0 | 11
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 3
Neurology-Other (Nervous system disorders) | 1 | 1 | 0 | 3
Neuropathy: motor (Nervous system disorders) | 3 | 2 | 0 | 1
Neuropathy: sensory (Nervous system disorders) | 27 | 13 | 0 | 20
Ocular/Visual-Other (Nervous system disorders) | 6 | 4 | 0 | 4
Pain - Head/headache (Nervous system disorders) | 55 | 7 | 0 | 24
Pain - Sinus (Nervous system disorders) | 4 | 0 | 0 | 3
Seizure (Nervous system disorders) | 0 | 2 | 0 | 2
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 0 | 0 | 0 | 2
Taste alteration (dysgeusia) (Nervous system disorders) | 6 | 1 | 0 | 2
Tremor (Nervous system disorders) | 2 | 0 | 0 | 6
Insomnia (Psychiatric disorders) | 26 | 6 | 0 | 11
Libido (Psychiatric disorders) | 1 | 1 | 0 | 2
Mood alteration - anxiety (Psychiatric disorders) | 31 | 5 | 0 | 8
Mood alteration - depression (Psychiatric disorders) | 15 | 7 | 0 | 11
Hemorrhage, GU - Urinary NOS (Renal and urinary disorders) | 1 | 0 | 0 | 2
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 2
Renal/Genitourinary-Other (Renal and urinary disorders) | 3 | 2 | 0 | 3
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 2
Gynecomastia (Reproductive system and breast disorders) | 0 | 1 | 0 | 3
Hemorrhage, GU - Vagina (Reproductive system and breast disorders) | 7 | 0 | 0 | 3
Pain - Pelvis (Reproductive system and breast disorders) | 1 | 0 | 0 | 2
Sexual/Reproductive Function-Other (Reproductive system and breast disorders) | 2 | 2 | 0 | 5
Vaginal dryness (Reproductive system and breast disorders) | 0 | 2 | 0 | 1
Vaginitis (not due to infection) (Reproductive system and breast disorders) | 0 | 0 | 0 | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 9 | 4 | 0 | 6
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 22 | 7 | 0 | 21
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 21 | 3 | 0 | 12
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 23 | 1 | 0 | 0
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0 | 4
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 8 | 3 | 0 | 6
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 11 | 2 | 0 | 6
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 2
Pulmonary/Upper Respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 9 | 4 | 0 | 6
Dermatology/Skin-Other (Skin and subcutaneous tissue disorders) | 11 | 2 | 0 | 9
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 8
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 21 | 1 | 0 | 4
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Nail changes (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 2
Pain - Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 3
Petechiae/purpura (hemorrhage into skin or mucosa) (Skin and subcutaneous tissue disorders) | 10 | 0 | 0 | 0
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 3
Pruritus/itching (Skin and subcutaneous tissue disorders) | 7 | 5 | 0 | 9
Rash/desquamation (Skin and subcutaneous tissue disorders) | 29 | 3 | 0 | 23
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 3 | 6 | 0 | 7
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 12 | 4 | 0 | 3
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 2
Flushing (Vascular disorders) | 4 | 0 | 0 | 4
Hot flashes/flushes (Vascular disorders) | 2 | 2 | 0 | 8
Hypertension (Vascular disorders) | 11 | 2 | 0 | 9
Hypotension (Vascular disorders) | 16 | 1 | 0 | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 12 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less